CLINICAL TRIAL: NCT00324103
Title: Antiretroviral Treatment With Structured Treatment Interruptions (STI) Versus Continuous Antiretroviral Treatment in HIV+ Patients With Persistent Suppression of Viral Replication
Brief Title: Structured Treatment Interruptions in Chronic HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS PART
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2006-05-10 (Estimated); Status verified 2005-10

CONDITIONS: HIV Infection
Keywords: HIV; Chronic Infection; Clinical Trial; Structured Treatment Interruption
MeSH Terms: conditions — HIV Infections; Persistent Infection

INTERVENTIONS:
Drug: Structured Treatment Interruptions

SUMMARY:
In the last years Structured Treatment Interruptions (STI) have been proposed to reduce HAART-related toxicity and to increase patients' compliance. ISS PART is a randomized comparison of repeated STIs versus continuous HAART in chronically HIV-infected subjects with persistent suppression of viral replication. The two arms of the study will be compared in terms of immunological response (proportion of patients with CD4>500/mmc) at 2 years.

DETAILED DESCRIPTION:
Patients are randomized in a 1 to 1 ratio to continue their current antiretroviral regimen (Arm A) or to undergo structured treatment interruptions (STI) (Arm B) according to the following scheme: STIs of 1, 1, 2, 2 and 3 months each followed by a 3-month therapy period.

During STIs, therapy is resumed in the presence of an HIV-RNA rebound > 50,000 copies/ml or of a CD4+ T cell decline > 25% of the baseline count (> 35% for patients with CD4+ > 500/mm3 at randomization). After the first cycle, subsequent STIs are performed only if an HIV-RNA level < 400 copies/ml is reached after 2 months of therapy resumption.

At the time of treatment interruptions patients in arm B who are on treatment with non-nucleoside reverse transcriptase inhibitors suspend these drugs first and continue the treatment with the other drugs of the combination for 3 days if nevirapine-treated and for 6 days in case of previous efavirenz-based regimen.

Patients are seen at the clinical site every three months for arm A and monthly for arm B. On these occasions, blood samples are obtained for biochemical and viro-immunological assessments.

The toxicity grading scale of the AIDS Clinical Trial Group (ACTG) is used for the reporting of clinical and laboratory adverse events.

In arm B, plasma genotype is obtained in samples taken after 15 or 30 days of drug suspension.

Patients will discontinue the study in case of : early therapy resumption for 2 consecutive times (only arm B patients); acute retroviral syndrome (only for arm B patients); AIDS-defining event; severe adverse event; pregnancy; non-compliance; patient' s request; physician's decision.

ELIGIBILITY:
Inclusion Criteria:

* first-line antiretroviral therapy (3 or 4 drugs) for 6 to 18 months (one previous therapy change for toxicity or non-compliance is allowed)
* HIV-RNA level below 400 copies/ml for at least 6 months;
* CD4+ count > 350 /mm3;
* pre-HAART CD4+ > 100/mm3
* no previous AIDS diagnosis.

Exclusion Criteria:

* Previous antiretroviral therapy with 1 or 2 drugs (except ARV prophylaxis in pregnancy)
* Pregnancy or breastfeeding
* Previous diagnosis of AIDS
* Grade 3 or 4 adverse event in the 15 days before enrolment
* Neoplasia
* Previous therapy with IL-2, interferon (in the last 2 years) or experimental therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-06; Study Completion 2004-06

PRIMARY OUTCOMES:
proportion of patients with CD4+ cell count above 500/mm3 at the end of follow-up (2 years) in the two treatment arms.

SECONDARY OUTCOMES:
occurrence of grade 3 or 4 adverse events (clinical and laboratory)
proportion of patients with HIV-RNA < 400 copies/ml at the end of follow-up
proportion of patients with CD4+ cell count > 350/mm3 at the end of follow-up
rate of virological failure
emergence of resistance
HIV-related events.

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Vella, MD, Study Chair — Istituto Superiore di Sanità
Locations (1):
- Istituto Superiore di Sanità, Rome, Italy